CLINICAL TRIAL: NCT04164992
Title: The Role of Endoscopic Ultrasound Radiofrequency Ablation (EUS RFA) in the Management of Not Resectable Pancreatic Cancer.
Brief Title: Endoscopic Ultrasound Radiofrequency Ablation (EUS-RFA) of Not-resectable Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Francesco Maria Di Matteo, MD; Head of Endoscopy department, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15/19
Record Dates: First submitted 2019-11-10; First posted 2019-11-15 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: endoscopic ultrasound radiofrequency ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- not resectable pancreatic cancer patients (Experimental): Patients with not-resectable pancreatic adenocarcinoma will be treated with endoscopic ultrasound radio frequency ablation
  Interventions: Device: EUSRA electrode needle connected to a radiofrequency generator (VIVA RF generator; STARmed, Seoul, S. Korea)

INTERVENTIONS:
Device: EUSRA electrode needle connected to a radiofrequency generator (VIVA RF generator; STARmed, Seoul, S. Korea) — The operative needle (EUSRA-STARMED) is a novel monopolar 18 gauge radiofrequency ablation (RFA) electrode that is placed in the echoendoscope operative channel. It is 140 cm long with a sharp conical 1 cm tip for energy delivery. The needle is associated with an internal cooling system connected via a pump to an external cold saline solution source (0 °C) that prevents the charring of the tip and improves the ablation accuracy.

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) remains one of the most aggressive tumors with a poor prognosis. Despite advancements in the multimodal approach, surgical resection still represents the only potentially curative treatment. However, more than 80% of patients are diagnosed at a non-resectable stage. Local ablative techniques are therefore emerging as complementary treatments in the multimodal strategy for un-resectable non-metastatic disease. Although radio frequency ablation (RFA) is already well established in other clinical settings, its role in the treatment of pancreatic lesions is still under evaluation. Several animal studies and small human clinical series are assessing the feasibility and safety of different RFA systems and settings to limit adverse events due to thermic damage, acute pancreatitis, stomach and duodenal transmural burns, perforations, and bleeding.

By now, three studies evaluated the feasibility and safety of EUS RFA in patients with locally advanced and metastatic PDAC showing that it is feasible and safe, However, the exact role of EUS-RFA in PDAC management must be further assessed.

The primary aim of this study is to evaluate the efficacy of endoscopic ultrasound radiofrequency ablation (EUS-RFA) by obtaining the tumour ablation in patients with locally advanced pancreatic cancer.

The secondary aim is to evaluate the safety of this procedure and its effect on symptoms.

Inclusion criteria: Patients with a cyto/histological diagnosis of PDAC, which was non-resectable and had no metastases after first line chemotherapy and/or radiotherapy; a solid pancreatic lesion that was resectable but not suitable for surgery due to the patient's comorbidities.

Patients enrolled will have a blood examination (including Carbohydrate Antigen 19.9) and a contrast-enhanced CT scan no more than 7 days before the procedure.

Patients will be administered a questionnaire about demographic features, symptoms, quality of life and drugs used. Tumours features and the type of chemotherapy protocol will also be recorded.

EUS-RFA will be performed with the patients placed on the le lateral position under deep sedation, employing a linear-array echoendoscope. An 19-gauge EUSRA electrode needle connected to a radiofrequency generator (VIVA RF generator; "STARmed", Seoul, S. Korea) will be used in all patients.

The procedure will be considered feasible if it will be possible to insert the electrode into the targeted point and to apply the radiofrequency energy for a sufficient time. All procedures will be started with a preset radiofrequency power of 30 Watt. If necessary, the procedure will be repeated by reinserting the needle in another part of the lesion until obtaining the largest possible ablation of the tumour.The radiofrequency power, duration of the ablation, the number of passages of the electrode necessary to obtain the ablation will be recorded.

Clinical evaluation and laboratory tests (complete blood count, liver function tests, and serum amylase/lipase levels) will be performed at 24 h after the procedure.

A contrast-enhanced computed tomography (CECT) scan will be performed one day and one month after the procedure to check the treatment outcome and exclude early and late adverse events.

Technical success will be defined by achieving tumour ablation defined by the presence of a hypodense area inside the tumour detectable at CECT scan. The volume of the ablated area (and its percentage in respect to the original tumour volume) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* cyto/histological diagnosis of PDAC, which was non-resectable and had no metastases after first line chemotherapy and/or radiotherapy (stage III);
* a solid pancreatic lesion that was resectable but not suitable for surgery or chemotherapy due to the patient's comorbidities:
* Performance status 0-1-2 (ECOG)

Exclusion Criteria:

* Age<18 anni
* Performance status > o = 3 (ECOG)
* Lesion not accessible with RFA needle
* Coagulation disorders
* Concomitant severe infections
* Pregnancy
* No informed consent given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Ablation efficacy of EUS-RFA | 1 month after the procedure
  Ablation efficacy of EUS-RF evaluated by changes of pancreatic tumor size (mm) at CE CT performed one months after the procedure.

SECONDARY OUTCOMES:
Number of post EUS-RFA adverse events | 24 hours after the procedure
  Post EUS RFA complications assessed with clinical evaluation (abdominal pain scored according with numerical rating scale (NRS), fever, vomit, stool blood) and biochemical exams (Hemoglobin, amylase, lipase, C-reactive protein).
Number of post EUS-RFA adverse events | 1 day and 1 month after the procedure.
  CE CT scan performed 1 day and 1 month after the procedure to exclude early and late adverse events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song TJ, Seo DW, Lakhtakia S, Reddy N, Oh DW, Park DH, Lee SS, Lee SK, Kim MH. Initial experience of EUS-guided radiofrequency ablation of unresectable pancreatic cancer. Gastrointest Endosc. 2016 Feb;83(2):440-3. doi: 10.1016/j.gie.2015.08.048. Epub 2015 Sep 4. PMID 26344883
- [Background] Scopelliti F, Pea A, Conigliaro R, Butturini G, Frigerio I, Regi P, Giardino A, Bertani H, Paini M, Pederzoli P, Girelli R. Technique, safety, and feasibility of EUS-guided radiofrequency ablation in unresectable pancreatic cancer. Surg Endosc. 2018 Sep;32(9):4022-4028. doi: 10.1007/s00464-018-6217-x. Epub 2018 May 15. PMID 29766302
- [Background] Crino SF, D'Onofrio M, Bernardoni L, Frulloni L, Iannelli M, Malleo G, Paiella S, Larghi A, Gabbrielli A. EUS-guided Radiofrequency Ablation (EUS-RFA) of Solid Pancreatic Neoplasm Using an 18-gauge Needle Electrode: Feasibility, Safety, and Technical Success. J Gastrointestin Liver Dis. 2018 Mar;27(1):67-72. doi: 10.15403/jgld.2014.1121.271.eus. PMID 29557417
- [Background] Kim HJ, Seo DW, Hassanuddin A, Kim SH, Chae HJ, Jang JW, Park DH, Lee SS, Lee SK, Kim MH. EUS-guided radiofrequency ablation of the porcine pancreas. Gastrointest Endosc. 2012 Nov;76(5):1039-43. doi: 10.1016/j.gie.2012.07.015. PMID 23078928